CLINICAL TRIAL: NCT06282978
Title: An Open Label, Multicenter, Phase II Study of Elranatamab as Single Agent for the Treatment of Relapsed or Refractory Myeloma in Patients Previously Exposed to Three-drug Classes (GEM-RANTAB)
Brief Title: Study of Elranatamab for Relapsed or Refractory Myeloma in Patients Previously Exposed to Three-drug Classes
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-RANTAB; 2023-504273-21 (EudraCT Number)
Record Dates: First submitted 2023-11-23; First posted 2024-02-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Relapsed Refractory Multiple Myeloma; Elranatamab
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: This is an open label, multicenter, phase II study of Elranatamab as single agent. The primary aiming is to evaluate the efficacy of elranatamab monotherapy in participants with relapsed refractory multiple myeloma (RRMM) who had received prior treatment with immunomodulatory drugs, protease inhibitors, and anti-CD38 therapy and were refractory to the last line of therapy as evaluated with the rate of complete Response and Undetectable Measurable Residual Disease. Efficacy refers to the rate of Undetectable Measurable Residual Disease at 6 and 12 months as per International Myeloma Working Group (IMWG) criteria evaluated by the investigators.
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Elranatamab (Experimental): Elranatamab will be administered by subcutaneous (SC) injection
  Interventions: Drug: Elranatamab (PF-06863135)

INTERVENTIONS:
Drug: Elranatamab (PF-06863135) — The scheme of administration includes weekly administrations for at least six 4-weeks cycles and, if patients have achieved at least PR (or better) persisting for at least 2 months, the dose interval should be changed from weekly to every other week. Treatment will be scheduled with a response-adapted duration and patients achieving undetectable measurable residual disease (MRD) and maintained for 12 months will stop therapy. After stopping therapy, and if the patient is in sustained undetectable MRD for at least 12 months, it would be possible to re-start treatment with elranatamab in case the MRD will be detectable or relapse from CR will occur. Patients who will not achieve undetectable MRD sustained for 12 months will receive continuous treatment until progressive disease.

SUMMARY:
The goal of this phase II, open-label, single-arm, multicenter study is to evaluate i) the efficacy and ii) safety of elranatamab monotherapy at the dose of 76 mg subcutaneously in participants with RRMM after at least one or two prior lines of therapy who have received prior treatment with immunomodulatory drugs, protease inhibitors, and anti-CD38 therapy and were refractory to the last line of therapy, defined as progression while receiving treatment or in the first 60 days after the last dose of treatment.

Efficacy refers to the rate of Undetectable Measurable Residual Disease at 6 and 12 months as per International Myeloma Working Group (IMWG) criteria evaluated by the investigators.

Safety refers to the measurement of:

i) Adverse events (AEs) and serious adverse events (SAEs) according to standard clinical and laboratory tests (hematology and chemistry, physical examination, vital sign measurements, and diagnostic tests).

ii) Incidence and severity of Cytokine Release Syndrome (CRS) and Immune effector cell associated neurotoxicity syndrome (ICANS) according to the American Society for Transplantation and Cellular Therapy (ASTCT) criteria.

iii) Incidence and severity of other neurotoxicities. iv) Incidence of cytopenias and infections

The study consists of a screening/baseline period, a treatment period, and a posttreatment follow-up period. The study includes a periodic review of safety data, that will be independently analyzed by the Data Safety Independent Committee (DSMC) and will recommend how to proceed with the study.

DETAILED DESCRIPTION:
Treatment with elranatamab will be initiated using a 2-step-up priming regimen: the initial doses of elranatamab will be 12 mg (Cycle 1 Day 1) and 32 mg (Cycle1 Day 4). Participants should be hospitalized and monitored for toxicity (especially CRS/ICANS) for at least 2 days (~48 hours) beginning on Cycle 1 Day 1, and for 1 day (~24 hours) for Cycle1 Day 4. The dose of elranatamab should be increased to 76 mg on Cycle 1 Day 8 as long as the participant meets the redosing criteria or deferred until the criteria are met.

The scheme of administration includes weekly administrations for at least six 4-weeks cycles and, if patients have achieved at least PR (or better) persisting for at least 2 months, the dose interval should be changed from weekly to every other week. Treatment will be scheduled with a response-adapted duration and patients achieving undetectable measurable residual disease and maintained for 12 months will stop therapy. After stopping therapy, and if the patient is in sustained undetectable measurable residual disease for at least 12 months, it would be possible to re-start treatment with elranatamab in case the measurable residual disease will be detectable or relapse from CR will occur. Patients who will not achieve undetectable measurable residual disease sustained for 12 months will receive continuous treatment until progressive disease. In both situations, the occurrence of unacceptable toxicity might result into the treatment discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years or older (at the time consent is obtained).
* Patient who, in the investigator's opinion, is able to comply with the protocol requirements.
* Prior diagnosis of MM as defined according to IMWG criteria.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Relapse multiple myeloma patients that have received at least 1 or 2 prior lines of therapy including at least to one proteasome inhibitor (bortezomib, carfilzomib or ixazomib), one immunomodulatory drug (lenalidomide is mandatory and patients can be also have been exposed to pomalidomide) and at least one anti-CD38 monoclonal antibody (daratumumab or isatuximab).
* Patients must be refractory to the last line of therapy, defined as progression while receiving treatment or in the first 60 days after the last dose of treatment.
* Patient must have a measurable secretory disease defined as either serum monoclonal protein of ≥ 0,5 g/dl or urine monoclonal (light chain) protein ≥ 200 mg/24 h. For patients in whom disease is only measurable by serum FLC, the involved FLC should be ≥ 10mg/dL (100 mg/L), with an abnormal serum FLC ratio.

Exclusion Criteria:

* Subject has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance (MGUS), smoldering multiple myeloma (SMM), POEMS syndrome (defined by the presence of peripheral neuropathy, organomegaly, endocrinopathy, monoclonal plasma-cells proliferative disorder, and skin changes) or plasma cell leukemia.
* Prior anti-BCMA treatment.
* Subject has peripheral neuropathy or neuropathic pain grade 2 or higher, as defined by the National Cancer Institute Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.
* History of Guillain-Barré syndrome (GBS) or GBS variants, or history of any Grade ≥3 peripheral motor polyneuropathy.
* Stem cell transplant within 12 weeks prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate the rate of Undetectable Measurable Residual Disease (uMRD) at 6 and 12 months as per International Myeloma Working Group (IMWG) criteria evaluated by the investigators of elranatamab in patients with relapsed/refractory multiple myeloma. | 5 Years
  To evaluate the rate of uMRD at 6 and 12 months (defined as the percentage of participants who are MRD negative by next generation flow cytometry (NGF) method and with a sensitivity level of at least 10-5) of elranatamab in patients with relapsed/refractory multiple myeloma. Next generation flow cytometry is a reproducible biomarker to detect the presence of phenotypically abnormal clonal plasma cells (Measurable Residual Disease). The presence of surface markers (CD138, CD27, CD38, CD56, CD45, CD19) and certain morphological characteristics (FSC and SSC) permit the specific identification of plasma cells (PC). This will permit unique, high specificity confirmation of the monoclonality of phenotypically abnormal plasma cells (by light chain restriction). Said cells will have been clearly identified by low antigen expression (CD19, CD27, CD38, CD45, CD81) or overexpression (CD56, CD117, CD138).

SECONDARY OUTCOMES:
To evaluate annually by NGF until loss of response, the rate of Undetectable Measurable Residual Disease (% of patients with MRD negative by NGF method and with a sensitivity level of 10-5) of elranatamab in patients with R/R multiple myeloma. | 5 Years
  To evaluate annually by Next Generation Flow Cytometry until loss of response, the rate of Undetectable Measurable Residual Disease (defined as the percentage of participants who are MRD negative by next generation flow cytometry method and with a sensitivity level of at least 10-5) of elranatamab in patients with relapsed/refractory multiple myeloma. Next generation flow cytometry is a reproducible biomarker to detect the presence of phenotypically abnormal clonal plasma cells (Measurable Residual Disease). The presence of surface markers (CD138, CD27, CD38, CD56, CD45, CD19) and certain morphological characteristics (FSC and SSC) permit the specific identification of plasma cells (PC). This will permit unique, high specificity confirmation of the monoclonality of phenotypically abnormal plasma cells (by light chain restriction). Said cells will have been clearly identified by low antigen expression (CD19, CD27, CD38, CD45, CD81) or overexpression (CD56, CD117, CD138).
Incidence and severity Adverse Events (AEs) and Serious Adverse Event (SAEs) as assessed by changes in laboratory values in blood and biochemistry tests. | 5 Years
  Blood test will measure complete blood count, hemoglobin, white blood cell count with differential count and platelet count.
  Biochemistry test will measure urea, creatinine, uric acid, bilirubin, alkaline phosphatase, LDH, AST, ALT, sodium, chloride, calcium, potassium and, glucose, magnesium, GGT, CRP and CPK.
Incidence and severity Adverse Events (AEs) and Serious Adverse Event (SAEs) as assessed by changes in physical examination and ECOG performance status scale (0-5). | 5 Years
  Physical examination will include the examination of general appearance, skin, neck (including thyroid), eyes, ears, nose, throat, lungs, heart, absomen, back, lymph nodes, extremities, vascular and neurological.
  Heght in centimetres (cm), body weight (kg).
  ECOG performance status has scale from 0 (fully active) to 5 (dead).
Incidence and severity Adverse Events (AEs) and Serious Adverse Event (SAEs) as assessed by changes in vital sign measurements. | 5 Years
  Vital signs will include the systolic and diastolic blood pressure, temperature, pulse rate, respiratory rate and oxygen saturation. Vital signs must be measured after resting for at least 5 minutes. Vital signs must be measured more frequently if warranted by the clinical condition of the participant. Vital signs are to be monitored at least every 4 hours (± 15 min) during first 48 hours after the first dose of study intervention (C1D1) and 24 hours after second dose of study intervention (C1D4).
Incidence and severity Adverse Events (AEs) and Serious Adverse Event (SAEs) as assessed by pregnancy test. | 5 Years
  Pregnancy test will be assessed by Serum beta-human chorionic gonadotropin (β -HCG) pregnancy test for female participants of childbearing potential only.
Incidence and severity Adverse Events (AEs) and Serious Adverse Event (SAEs) as assessed by changes in 12-lead ECG. | 5 Years
  Electrocardiograms (ECG) must be recorded after 10 minutes rest in the supine position to ensure a table baseline. ECG will be performed at screening and end of treatment, but this test can be repeated throughout the study at the discretion of investigators.
  A standard 12-lead ECG will include a general diagnostic impression as well as measurement of the heart rate, PR interval, QRS duration, QT interval, and the Fridericia-corrected QT interval (QTcF). The QTcF must be used for clinical decisions. The investigator must calculate QTcF if its is not auto calculated by the ECG machine.
Incidence and severity Adverse Events (AEs) and Serious Adverse Event (SAEs) as assessed by changes in Echocardiogram / MUGA. | 5 Years
  This test will be will be performed at screening and end of treatment, but can be repeated when clinically indicated based on patient condition. A MUGA scan is also valid.
  Echocardiogram will include a Left ventricular ejection fraction (LVEF %).
To determine Circulating Tumor Cells (CTC) at baseline to evaluate its prognostic value. | 5 Years
  Counting of CTC by next generation flow cytometry and correlation of the number of CTC with MRD and survival will be done.
To determine serum BCMA levels and its correlation with response. | 5 Years
  Values of BCMA in blood samples (serum) will be correlated with MRD and survival.
To do gene expression techniques (RNA sequencing and single cell sequencing studies) coupled with intelligent clinical and molecular data analysis (i.e. machine learning) to identify factors that could predict response to elranatamab. | 5 Years
  Statistical analysis will be done to find significant changes in gene expression which identify markers of response (MRD negativity or positivity) to elranatamab.
To determine MRD value with alternative methods | 5 Years
  Mass spectrometry (alternative method) will be used to complement the evaluation of the response by the conventional techniques like electrophoresis, immunofixation and next generation flow cytometry.
To characterize patients' immune system | 5 Years
  Next generation flow cytometry (NGF) will be used to identify and characterize T, B, NK, monocytes and normal/clonal Plasma Cells (including BCMA antigen expression).
  NGF for the quantification of soluble factors: IL6, IL2, IFNγ and TNFα.
To define genomic determinants of response/resistance | 5 Years
  This determination will be done by next generation flow cytometry by Fluorescence-Activated Cell Sorting (FACS) sorting of T and Pathological Plasma Cells at inclusion and at progressive disease, and of T cells after the first dose.
To evaluate Overall Response Rate of elranatamab in patients with relapsed/refractory multiple myeloma. | 5 years
  Measurement of Overall response rate and the different responses categories according to the IMWG criteria as evaluated by investigator
To evaluate Duration of Response of elranatamab in patients with relapsed/refractory multiple myeloma. | 5 years
  Duration of response refers to the time from Complete Remission achievement to loss of response/disease progression.
To evaluate Time to first and best response of elranatamab in patients with relapsed/refractory multiple myeloma. | 5 years
  Time to first and best response refers to the time from first Complete Remission achievement to disease progression. The degree of response is also assessed and correltaes with the level of MRD measured by Next Generation Flow Cytometry.
To evaluate Progression-free survival (PFS) of elranatamab in patients with relapsed/refractory multiple myeloma. | 5 years
  PFS is defined as the time from the date of first dose of study drug to the date of first documented disease progression, as defined in the International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurs first. For subjects who have not progressed and are alive, data will be censored at the last disease evaluation before the start of any subsequent anti-myeloma therapy. PFS is measured in months
To evaluate Overall survival (OS) of elranatamab in patients with relapsed/refractory multiple myeloma. | 5 years
  OS is defined as the time from the date of first dose of study drug to the date of the subject's death. If the subject is alive or the vital status is unknown, then the subject's data will be censored at the date the subject was last known to be alive. OS is measured in months.
To evaluate PFS in those patients who stop treatment because of sustained MRD-positive for 12 months of elranatamab in patients with relapsed/refractory multiple myeloma. | 5 yerars
  The same definitions used above but restricted to patients with poor response to therapy (sustained MRD-positive for 12 months)
To evaluate OS in those patients who stop treatment because of sustained MRD-positive for 12 months of elranatamab in patients with relapsed/refractory multiple myeloma. | 5 yerars
  The same definitions used above but restricted to patients with poor response to therapy (sustained MRD-positive for 12 months)
To evaluate the Incidence of neurologic effects related to elranatamab in patients with relapsed/refractory multiple myeloma. | 5 years
  Incidence and severity of Cytokine Release Syndrome (CRS) and Immune effector cell associated neurotoxicity syndrome (ICANS) will be collected according to the American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Incidence and degree of other neurotoxicities.
To evaluate the Incidence of cytopenias and infections related to elranatamab in patients with relapsed/refractory multiple myeloma. | 5 years
  Incidence and degree of cytopenias and infections according to the American Society for Transplantation and Cellular Therapy (ASTCT) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: María-Victoria Mateos, MD, Study Chair — University of Salamanca
Locations (15):
- Spain (15):
  - Hospital Clínico Universitario de Santiago ~ CHUS, Santiago de Compostela, A Coruña
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Institut Catala d'Oncologia (ICO) Badalona - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Institut Catala d'Oncologia (ICO) Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - CHU de Gran Canaria Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital HM Sanchinarro, PAU de Sanchinarro, Madrid
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Clinica Universidad Navarra (CUN), Pamplona, Navarre
  - H. Clínic i Provincial de Barcelona, Barcelona
  - Hospital de Cabueñes, Gijón
  - Instituto de Investigación Sanitaria Hospital 12 de Octubre, Madrid
  - Hospital Clínico Universitario Salamanca, Salamanca
  - C.H. de Toledo (Virgen de la Salud), Toledo

IPD SHARING:
Plan to Share IPD: No
All participant data relating to the study will be recorded on electronic CRF unless transmitted to the sponsor or designee electronically (e.g., laboratory data). The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the eCRF. Results of this clinical trial, positive or negative, will be presented at scientific conferences and published in scientific journals.

REFERENCES:
- [Background] van de Donk NWCJ, Pawlyn C, Yong KL. Multiple myeloma. Lancet. 2021 Jan 30;397(10272):410-427. doi: 10.1016/S0140-6736(21)00135-5. PMID 33516340
- [Background] Dimopoulos MA, Moreau P, Terpos E, Mateos MV, Zweegman S, Cook G, Delforge M, Hajek R, Schjesvold F, Cavo M, Goldschmidt H, Facon T, Einsele H, Boccadoro M, San-Miguel J, Sonneveld P, Mey U; EHA Guidelines Committee. Electronic address: guidelines@ehaweb.org; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. Multiple myeloma: EHA-ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-updagger. Ann Oncol. 2021 Mar;32(3):309-322. doi: 10.1016/j.annonc.2020.11.014. Epub 2021 Feb 3. No abstract available. PMID 33549387
- [Background] Moreau P, Kumar SK, San Miguel J, Davies F, Zamagni E, Bahlis N, Ludwig H, Mikhael J, Terpos E, Schjesvold F, Martin T, Yong K, Durie BGM, Facon T, Jurczyszyn A, Sidana S, Raje N, van de Donk N, Lonial S, Cavo M, Kristinsson SY, Lentzsch S, Hajek R, Anderson KC, Joao C, Einsele H, Sonneveld P, Engelhardt M, Fonseca R, Vangsted A, Weisel K, Baz R, Hungria V, Berdeja JG, Leal da Costa F, Maiolino A, Waage A, Vesole DH, Ocio EM, Quach H, Driessen C, Blade J, Leleu X, Riva E, Bergsagel PL, Hou J, Chng WJ, Mellqvist UH, Dytfeld D, Harousseau JL, Goldschmidt H, Laubach J, Munshi NC, Gay F, Beksac M, Costa LJ, Kaiser M, Hari P, Boccadoro M, Usmani SZ, Zweegman S, Holstein S, Sezer O, Harrison S, Nahi H, Cook G, Mateos MV, Rajkumar SV, Dimopoulos MA, Richardson PG. Treatment of relapsed and refractory multiple myeloma: recommendations from the International Myeloma Working Group. Lancet Oncol. 2021 Mar;22(3):e105-e118. doi: 10.1016/S1470-2045(20)30756-7. PMID 33662288
- [Background] Casanova M, Mateos MV, de Arriba F, al. e. Determination of the Value Contribution of Belantamab Mafodotin (Belamaf; BLENREP®) for the Treatment of Triple-Class Refractory Multiple Myeloma in Spain through Reflective Multi-Criteria Decision Analysis. Rev Esp Econ Salud. 2021;16(3):58-69.
- [Background] European Medicines Agency. NEXPOVIO. Summary of Product Characteristics. Available at: https://www.ema.europa.eu/en/documents/product-information/nexpovio-epar-product-informat ion_es.pdf . 2022.
- [Background] European Medicines Agency. BLENREP. Summary of Product Characteristics. Available at: https://www.ema.europa.eu/en/documents/product-information/blenrep-epar-product-informa tion_es.pdf . 2022.
- [Background] Yang Q, Li X, Zhang F, Yang Q, Zhou W, Liu J. Efficacy and Safety of CAR-T Therapy for Relapse or Refractory Multiple Myeloma: A systematic review and meta-analysis. Int J Med Sci. 2021 Feb 18;18(8):1786-1797. doi: 10.7150/ijms.46811. eCollection 2021. PMID 33746596
- [Background] Zhang L, Shen X, Yu W, Li J, Zhang J, Zhang R, Li J, Chen L. Comprehensive meta-analysis of anti-BCMA chimeric antigen receptor T-cell therapy in relapsed or refractory multiple myeloma. Ann Med. 2021 Dec;53(1):1547-1559. doi: 10.1080/07853890.2021.1970218. PMID 34459681
- [Background] Cho SF, Yeh TJ, Anderson KC, Tai YT. Bispecific antibodies in multiple myeloma treatment: A journey in progress. Front Oncol. 2022 Oct 18;12:1032775. doi: 10.3389/fonc.2022.1032775. eCollection 2022. PMID 36330495
- [Background] Food and Drug Administration. FDA approves idecabtagene vicleucel for multiple myeloma. Available at: https://www.fda.gov/drugs/resources-information-approved-drugs/fda-approves-idecabtagenevicleucel- multiple-myeloma . 2022.
- [Background] European Medicines Agency. Abecma. Summary of Product Characteristics. Available at: https://www.ema.europa.eu/en/documents/product-information/abecma-epar-product-informati on_en.pdf . 2022.
- [Background] Food and Drug Administration. FDA approves ciltacabtagene autoleucel for relapsed or refractory multiple myeloma. Available at: https://www.fda.gov/drugs/resources-information-approved-drugs/fda-approves-ciltacabtageneautoleucel- relapsed-or-refractory-multiple-myeloma . 2022.
- [Background] European Medicines Agency. CARVYKTI. Summary of Product Characteristics. Available at: https://www.ema.europa.eu/en/documents/product-information/carvykti-epar-product-informatio n_en.pdf . 2022.
- [Background] Munshi NC, Anderson LD Jr, Shah N, Madduri D, Berdeja J, Lonial S, Raje N, Lin Y, Siegel D, Oriol A, Moreau P, Yakoub-Agha I, Delforge M, Cavo M, Einsele H, Goldschmidt H, Weisel K, Rambaldi A, Reece D, Petrocca F, Massaro M, Connarn JN, Kaiser S, Patel P, Huang L, Campbell TB, Hege K, San-Miguel J. Idecabtagene Vicleucel in Relapsed and Refractory Multiple Myeloma. N Engl J Med. 2021 Feb 25;384(8):705-716. doi: 10.1056/NEJMoa2024850. PMID 33626253
- [Background] Berdeja JG, Madduri D, Usmani SZ, Jakubowiak A, Agha M, Cohen AD, Stewart AK, Hari P, Htut M, Lesokhin A, Deol A, Munshi NC, O'Donnell E, Avigan D, Singh I, Zudaire E, Yeh TM, Allred AJ, Olyslager Y, Banerjee A, Jackson CC, Goldberg JD, Schecter JM, Deraedt W, Zhuang SH, Infante J, Geng D, Wu X, Carrasco-Alfonso MJ, Akram M, Hossain F, Rizvi S, Fan F, Lin Y, Martin T, Jagannath S. Ciltacabtagene autoleucel, a B-cell maturation antigen-directed chimeric antigen receptor T-cell therapy in patients with relapsed or refractory multiple myeloma (CARTITUDE-1): a phase 1b/2 open-label study. Lancet. 2021 Jul 24;398(10297):314-324. doi: 10.1016/S0140-6736(21)00933-8. Epub 2021 Jun 24. PMID 34175021
- [Background] Food and Drug Administration. FDA approves teclistamab-cqyv for relapsed or refractory multiple myeloma. Available at: https://www.fda.gov/drugs/resources-information-approved-drugs/fda-approves-teclistamab-cq yv-relapsed-or-refractory-multiple-myeloma . 2022.
- [Background] European Medicines Agency. TECVAYLI. Summary of Product Characteristics. Available at: https://www.ema.europa.eu/en/documents/product-information/tecvayli-epar-product-informatio n_en.pdf . 2022.
- [Background] Moreau P, Garfall AL, van de Donk NWCJ, Nahi H, San-Miguel JF, Oriol A, Nooka AK, Martin T, Rosinol L, Chari A, Karlin L, Benboubker L, Mateos MV, Bahlis N, Popat R, Besemer B, Martinez-Lopez J, Sidana S, Delforge M, Pei L, Trancucci D, Verona R, Girgis S, Lin SXW, Olyslager Y, Jaffe M, Uhlar C, Stephenson T, Van Rampelbergh R, Banerjee A, Goldberg JD, Kobos R, Krishnan A, Usmani SZ. Teclistamab in Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2022 Aug 11;387(6):495-505. doi: 10.1056/NEJMoa2203478. Epub 2022 Jun 5. PMID 35661166
- [Background] Lassiter G, Bergeron C, Guedry R, Cucarola J, Kaye AM, Cornett EM, Kaye AD, Varrassi G, Viswanath O, Urits I. Belantamab Mafodotin to Treat Multiple Myeloma: A Comprehensive Review of Disease, Drug Efficacy and Side Effects. Curr Oncol. 2021 Jan 21;28(1):640-660. doi: 10.3390/curroncol28010063. PMID 33494319
- [Background] Tai YT, Anderson KC. Targeting B-cell maturation antigen in multiple myeloma. Immunotherapy. 2015;7(11):1187-99. doi: 10.2217/imt.15.77. Epub 2015 Sep 15. PMID 26370838
- [Background] Tai YT, Li XF, Breitkreutz I, Song W, Neri P, Catley L, Podar K, Hideshima T, Chauhan D, Raje N, Schlossman R, Richardson P, Munshi NC, Anderson KC. Role of B-cell-activating factor in adhesion and growth of human multiple myeloma cells in the bone marrow microenvironment. Cancer Res. 2006 Jul 1;66(13):6675-82. doi: 10.1158/0008-5472.CAN-06-0190. PMID 16818641
- [Background] Sanchez E, Li M, Kitto A, Li J, Wang CS, Kirk DT, Yellin O, Nichols CM, Dreyer MP, Ahles CP, Robinson A, Madden E, Waterman GN, Swift RA, Bonavida B, Boccia R, Vescio RA, Crowley J, Chen H, Berenson JR. Serum B-cell maturation antigen is elevated in multiple myeloma and correlates with disease status and survival. Br J Haematol. 2012 Sep;158(6):727-38. doi: 10.1111/j.1365-2141.2012.09241.x. Epub 2012 Jul 18. PMID 22804669
- [Background] Novak AJ, Darce JR, Arendt BK, Harder B, Henderson K, Kindsvogel W, Gross JA, Greipp PR, Jelinek DF. Expression of BCMA, TACI, and BAFF-R in multiple myeloma: a mechanism for growth and survival. Blood. 2004 Jan 15;103(2):689-94. doi: 10.1182/blood-2003-06-2043. Epub 2003 Sep 25. PMID 14512299
- [Background] Shah N, Chari A, Scott E, Mezzi K, Usmani SZ. B-cell maturation antigen (BCMA) in multiple myeloma: rationale for targeting and current therapeutic approaches. Leukemia. 2020 Apr;34(4):985-1005. doi: 10.1038/s41375-020-0734-z. Epub 2020 Feb 13. PMID 32055000
- [Background] Lesokhin AM, Raje N, Gasparetto CJ, et al. A Phase I, Open-Label Study to Evaluate the Safety, Pharmacokinetic, Pharmacodynamic, and Clinical Activity of PF-06863135, a B-Cell Maturation Antigen/CD3 Bispecific Antibody, in Patients with Relapsed/Refractory Advanced Multiple Myeloma. Blood. 2018;132(Supplement 1):3229-3229.
- [Background] Panowski SH, Kuo TC, Zhang Y, Chen A, Geng T, Aschenbrenner L, Kamperschroer C, Pascua E, Chen W, Delaria K, Farias S, Bateman M, Dushin RG, Chin SM, Van Blarcom TJ, Yeung YA, Lindquist KC, Chunyk AG, Kuang B, Han B, Mirsky M, Pardo I, Buetow B, Martin TG, Wolf JL, Shelton D, Rajpal A, Strop P, Chaparro-Riggers J, Sasu BJ. Preclinical Efficacy and Safety Comparison of CD3 Bispecific and ADC Modalities Targeting BCMA for the Treatment of Multiple Myeloma. Mol Cancer Ther. 2019 Nov;18(11):2008-2020. doi: 10.1158/1535-7163.MCT-19-0007. Epub 2019 Aug 21. PMID 31434693
- [Background] Karwacz K, Hooper AT, Chang C-PB, et al. Abstract 4557: BCMA-CD3 bispecific antibody PF-06863135: Preclinical rationale for therapeutic combinations. Immunology. 2020;80:4557-4557.
- [Background] Sebag M, Raje NS, Bahlis NJ, et al. Elranatamab (PF-06863135), a B-Cell Maturation Antigen (BCMA) Targeted CD3-Engaging Bispecific Molecule, for Patients with Relapsed or Refractory Multiple Myeloma: Results from Magnetismm-1. Blood. 2021;138(Supplement 1):895-895
- [Background] Raje N, Bahlis NJ, Costello C, al. e. Elranatamab, a BCMA Targeted T-Cell Engaging Bispecific Antibody, Induces Durable Clinical and Molecular Responses for Patients with Relapsed or Refractory Multiple Myeloma. Blood. 2022;140:388-390.
- [Background] Lesokhin AM, Arnulf B, Niesvizky R, et al. Initial safety results for MagnetisMM-3: A phase 2 trial of elranatamab, a B-cell maturation antigen (BCMA)-CD3 bispecific antibody, in patients (pts) with relapsed/refractory (R/R) multiple myeloma (MM). Journal of Clinical Oncology. 2022;40(16_suppl):8006-8006.
- [Background] Bahlis NJ, Tomasson MH, Mohty M, al. e. Efficacy and Safety of Elranatamab in Patients with Relapsed/Refractory Multiple Myeloma Naïve to B-Cell Maturation Antigen (BCMA)-Directed Therapies: Results from Cohort a of the Magnetismm-3 Study. Blood. 2022;140:391-393.
- [Background] Pfizer. Pfizer Presents Updated Favorable Elranatamab Data from Pivotal Phase 2 MagnetisMM-3 Trial. Press release available at: https://www.pfizer.com/news/press-release/press-release-detail/pfizer-presents-updated-favora ble-elranatamab-data-pivotal . 2022.
- [Background] Pfizer. PF-06863135 As Single Agent And In Combination With Immunomodulatory Agents In Relapse/Refractory Multiple Myeloma. ClinicalTrials.gov Identifier: NCT03269136. Updated July 11, 2022. Accessed September 17, 2022. https://clinicaltrials.gov/ct2/show/NCT03269136 . 2022.
- [Background] Pfizer. Pfizer Presents First Data from Planned Interim Analysis of Pivotal Phase 2 MagnetisMM-3 Trial of BCMA-CD3 Bispecific Antibody Elranatamab Under Investigation for Relapsed/Refractory Multiple Myeloma. Press release available at: https://www.pfizer.com/news/press-release/press-release-detail/pfizer-presents-first-data-plann ed-interim-analysis-pivotal . 2022.
- [Background] Elmeliegy M, Viqueira A, Erik Vandendries E, al. e. Dose Optimization to Mitigate the Risk of CRS with Elranatamab in Multiple Myeloma. Presented at the: 64th ASH Annual Meeting & Exposition, New Orleans, December 10-13, 2022. Available at: https://ash.confex.com/ash/2022/webprogram/Paper169971.html . 2022.
- [Background] Munshi NC, Avet-Loiseau H, Rawstron AC, Owen RG, Child JA, Thakurta A, Sherrington P, Samur MK, Georgieva A, Anderson KC, Gregory WM. Association of Minimal Residual Disease With Superior Survival Outcomes in Patients With Multiple Myeloma: A Meta-analysis. JAMA Oncol. 2017 Jan 1;3(1):28-35. doi: 10.1001/jamaoncol.2016.3160. PMID 27632282
- [Background] Lahuerta JJ, Paiva B, Vidriales MB, Cordon L, Cedena MT, Puig N, Martinez-Lopez J, Rosinol L, Gutierrez NC, Martin-Ramos ML, Oriol A, Teruel AI, Echeveste MA, de Paz R, de Arriba F, Hernandez MT, Palomera L, Martinez R, Martin A, Alegre A, De la Rubia J, Orfao A, Mateos MV, Blade J, San-Miguel JF; GEM (Grupo Espanol de Mieloma)/PETHEMA (Programa para el Estudio de la Terapeutica en Hemopatias Malignas) Cooperative Study Group. Depth of Response in Multiple Myeloma: A Pooled Analysis of Three PETHEMA/GEM Clinical Trials. J Clin Oncol. 2017 Sep 1;35(25):2900-2910. doi: 10.1200/JCO.2016.69.2517. Epub 2017 May 12. PMID 28498784
- [Background] Carson JL, Guyatt G, Heddle NM, Grossman BJ, Cohn CS, Fung MK, Gernsheimer T, Holcomb JB, Kaplan LJ, Katz LM, Peterson N, Ramsey G, Rao SV, Roback JD, Shander A, Tobian AA. Clinical Practice Guidelines From the AABB: Red Blood Cell Transfusion Thresholds and Storage. JAMA. 2016 Nov 15;316(19):2025-2035. doi: 10.1001/jama.2016.9185. PMID 27732721
- [Background] Kumar SK, Callander NS, Adekola K, Anderson L, Baljevic M, Campagnaro E, Castillo JJ, Chandler JC, Costello C, Efebera Y, Faiman M, Garfall A, Godby K, Hillengass J, Holmberg L, Htut M, Huff CA, Kang Y, Hultcrantz M, Larson S, Liedtke M, Martin T, Omel J, Shain K, Sborov D, Stockerl-Goldstein K, Weber D, Keller J, Kumar R. Multiple Myeloma, Version 3.2021, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2020 Dec 2;18(12):1685-1717. doi: 10.6004/jnccn.2020.0057. PMID 33285522
- [Background] Raje NS, Anaissie E, Kumar SK, Lonial S, Martin T, Gertz MA, Krishnan A, Hari P, Ludwig H, O'Donnell E, Yee A, Kaufman JL, Cohen AD, Garderet L, Wechalekar AF, Terpos E, Khatry N, Niesvizky R, Yi Q, Joshua DE, Saikia T, Leung N, Engelhardt M, Mothy M, Branagan A, Chari A, Reiman AJ, Lipe B, Richter J, Rajkumar SV, Miguel JS, Anderson KC, Stadtmauer EA, Prabhala RH, McCarthy PL, Munshi NC. Consensus guidelines and recommendations for infection prevention in multiple myeloma: a report from the International Myeloma Working Group. Lancet Haematol. 2022 Feb;9(2):e143-e161. doi: 10.1016/S2352-3026(21)00283-0. PMID 35114152
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Richardson PG, Delforge M, Beksac M, Wen P, Jongen JL, Sezer O, Terpos E, Munshi N, Palumbo A, Rajkumar SV, Harousseau JL, Moreau P, Avet-Loiseau H, Lee JH, Cavo M, Merlini G, Voorhees P, Chng WJ, Mazumder A, Usmani S, Einsele H, Comenzo R, Orlowski R, Vesole D, Lahuerta JJ, Niesvizky R, Siegel D, Mateos MV, Dimopoulos M, Lonial S, Jagannath S, Blade J, Miguel JS, Morgan G, Anderson KC, Durie BG, Sonneveld P. Management of treatment-emergent peripheral neuropathy in multiple myeloma. Leukemia. 2012 Apr;26(4):595-608. doi: 10.1038/leu.2011.346. Epub 2011 Dec 23. PMID 22193964
- [Background] Topp MS, Duell J, Zugmaier G, Attal M, Moreau P, Langer C, Kronke J, Facon T, Salnikov AV, Lesley R, Beutner K, Kalabus J, Rasmussen E, Riemann K, Minella AC, Munzert G, Einsele H. Anti-B-Cell Maturation Antigen BiTE Molecule AMG 420 Induces Responses in Multiple Myeloma. J Clin Oncol. 2020 Mar 10;38(8):775-783. doi: 10.1200/JCO.19.02657. Epub 2020 Jan 2. PMID 31895611